CLINICAL TRIAL: NCT01703299
Title: Emergence of Resistance in Intestinal Microflora During Carbapenem Treatments
Acronym: ERIC
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: CRC11016
Record Dates: First submitted 2012-09-25; First posted 2012-10-10 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2014-06

CONDITIONS: Carbapenem-induced Resistance
Keywords: imipenem; ertapenem; resistance; commensal flora

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — faeces, bacterial DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- imipenem-treated patients: imipenem-treated patients
- ertapenem-treated patients: ertapenem-treated patients

SUMMARY:
The use of carbapenems, very broad spectrum antibiotics of last resort, is becoming more common due to the increased prevalence in the hospital and community of extended spectrum β-lactamase (ESBL) producing gram-negative bacilli (GNB), including CTX-M type, which are resistant to all other β-lactam antibiotics. Meanwhile, it creates a selective pressure towards emergence of strains which are also resistant to carbapenems, placing patients in a catastrophic situation of therapeutic dead-end. A better understanding of the mechanisms of emergence of BGN resistant to carbapenems is necessary to optimize their use and undertake preventive measures to preserve their effectiveness. The aim of the study is to evaluate and describe the emergence of carbapenem-induced resistant GNB in patient intestinal microflora.

DETAILED DESCRIPTION:
The use of carbapenems, very broad spectrum antibiotics of last resort, is becoming more common due to the increased prevalence in the hospital and community of extended spectrum β-lactamase (ESBL) producing gram-negative bacilli (GNB), including CTX-M type, which are resistant to all other β-lactam antibiotics. Meanwhile, it creates a selective pressure towards emergence of strains which are also resistant to carbapenems, placing patients in a catastrophic situation of therapeutic dead-end. A better understanding of the mechanisms of emergence of BGN resistant to carbapenems is necessary to optimize their use and undertake preventive measures to preserve their effectiveness.

Hypotheses: Carbapenems induce in treated patients the emergence of resistant GNB in intestinal flora and have an impact on colonization resistance of the gut microbiota.

Primary objective: To determine the frequency of emergence of carbapenems resistant GNB in the intestinal flora at the end of a treatment by imipenem or ertapenem.

Secondary objective(s):

* Assess the presence of carbapenem resistant GNB in the intestinal flora before treatment.
* Evaluate the presence and / or persistence of carbapenem resistant GNB in the intestinal flora on day 3 of treatment, and 15 days and 1 month after the end of treatment.
* Determine the molecular mechanisms of resistance of strains of interest.
* Describe the gastrointestinal tract colonization by non-commensal microorganisms before and after treatment (impact on colonization resistance).
* Describe the characteristics of patients with emergence of resistance compared to patients who do not.
* Proper conservation of stool of 10 patients for metagenomic and/or metatranscriptomic analysis of changes in the intestinal flora.

Primary endpoint: Presence of carbapenem resistant GNB in the stool at the end of treatment in patients who did not before, after culture on selective media.

Secondary endpoints:

* Presence of carbapenem resistant GNB in stools before treatment, at day 3 and 15 days and 1 month after stopping treatment, after culture on selective media.
* PCR and sequencing of resistance genes from strains of interest.
* Colonization of the digestive tract by non-commensal microorganisms before and after treatment.
* Characteristics of patients with or without emergence of resistance.

ELIGIBILITY:
Inclusion Criteria:

* age> or = 18 years old
* hospitalized
* initiating a treatment by imipenem or ertapenem-
* faeces harvested before the beginning of treatment
* written informed consent from the patient or from a relative if the patient is incapable of expressing his/her consent
* reachable by phone after hospitalization (only for patients able to express their consent).

Exclusion Criteria :

* hospitalized in intensive care unit
* concomitant antibiotic treatment (except aminosid or vancomycin for less than 4 days).

Secondary exclusion criteria :

* introduction of other antibiotics during carbapenem treatment (except vancomycin or aminosid)
* vancomycin treatment for more than 4 days during carbapenem treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospitalized patients initiating a carbapenem treatment
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
presence of carbapenem-resistant gram-negative bacteria at the end of carbapenem treatment in faeces of patients who were free of carbapenem-resistant gram-negative bacteria before the beginning of treatment | at the end of carbapenem treatment period which usually lasts between 2 and 15 days
  faecal bacterial growth on selective culture media

SECONDARY OUTCOMES:
presence of carbapenem-resistant gram-negative bacteria in patient faeces before carbapenem treatment, at day 3 of carbapenem treatment and at day 15 et day 30 after the end of carbapenem treatment | before, at day 3 of carbapenem treatment and at day 15 and day 30 after the end of carbapenem treatment
  faecal bacterial growth on selective culture media

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Andremont, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (5):
- France (5):
  - Hôpital Beaujon, Clichy
  - Hôpital Louis Mourier, Colombes
  - Hôpital Bichat-Claude Bernard, Paris
  - Hôpital Saint-Louis, Paris
  - Hôpital Paul Brousse, Villejuif

REFERENCES:
- [Derived] Grall N, Lazarevic V, Gaia N, Couffignal C, Laouenan C, Ilic-Habensus E, Wieder I, Plesiat P, Angebault C, Bougnoux ME, Armand-Lefevre L, Andremont A, Duval X, Schrenzel J. Unexpected persistence of extended-spectrum beta-lactamase-producing Enterobacteriaceae in the faecal microbiota of hospitalised patients treated with imipenem. Int J Antimicrob Agents. 2017 Jul;50(1):81-87. doi: 10.1016/j.ijantimicag.2017.02.018. Epub 2017 May 10. PMID 28499958